CLINICAL TRIAL: NCT04297124
Title: A Phase 1, Single-Center, Open-Label Study, to Evaluate the Metabolism and Excretion of [14C]-CC-90009 in Healthy Male Subjects
Brief Title: A Study to Evaluate the Metabolism and Excretion of [14C]-CC-90009 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-90009-CP-001; U1111-1248-0508 (Other: WHO)
Record Dates: First submitted 2020-03-04; First posted 2020-03-05 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Healthy Volunteer
Keywords: CC-90009; Metabolism; Healthy Male
MeSH Terms: interventions — CC-90009

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C]-CC-90009 (Experimental): A single IV dose of 0.6 mg [14C]-CC-90009 containing approximately 2 µCi of radioactivity will be administered on Day 1 under fasted conditions.
  Interventions: Drug: CC-90009; Radiation: [14C]

INTERVENTIONS:
Drug: CC-90009 — 0.6 mg [ 14C]-CC-90009 administered IV as a single dose
Radiation: [14C] — A single dose of [ 14C]-CC-90009 will contain approximately 2 µCi of radioactivity.

SUMMARY:
CC-90009-CP-001 is a Phase 1, single-center, open-label, clinical pharmacology study to measure how much CC 90009 gets into the bloodstream, how much is eliminated in urine and stool, and how long it takes the body to get rid of it. In addition, the safety and tolerability of CC 90009 will be evaluated.

DETAILED DESCRIPTION:
The primary objective of the study is to characterize the biotransformation and excretion of [14C]-CC-90009 following a single intravenous (IV) dose of 0.6 mg [14C]-CC-90009 in healthy male subjects. The secondary objective of the study is to evaluate the safety and tolerability. The total radioactivity of [14C]-CC-90009 will be 2 μCi.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Subject is ≥ 18 and ≤ 55 years of age at the time of signing the informed consent form (ICF).
2. Subject is male.
3. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
4. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.
5. Subject is in good health, as determined by the Investigator based on a physical examination at screening.
6. Subject agrees to abide by the requirements and restrictions outlined in the CC-90009 Pregnancy Prevention Plan for Subjects in Clinical Trials.
7. All subjects must avoid donating semen or sperm and practice complete abstinence (True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence [eg calendar, ovulation, symptothermal or post ovulation methods] and withdrawal are not acceptable methods of contraception.) or condom use during sexual contact with a pregnant female or a female of childbearing potential (FCBP) while receiving CC-90009 and for at least 28 days after the dose, even if he has undergone a successful vasectomy. If engaging in sexual contact, inform their partners who are FCBP to use two methods of reliable contraception, one highly effective and one additional effective, throughout the entire duration of CC-90009 and for at least 28 days after their dose of CC-90009. Partners of male subjects who are females of childbearing potential must use contraception during the same duration as the male subject to avoid pregnancy. If a pregnancy occurs with your partner, notify the doctor conducting the study immediately. The following are examples of highly effective and additional effective methods of contraception:

   * Examples of highly effective methods:

     * Intrauterine device (IUD)
     * Hormonal (birth control pills, injections, implants, levonorgestrel-releasing intrauterine system [IUS], medroxyprogesterone acetate depot injections, ovulation inhibitory progesterone-only pills [e.g. desogestrel])
     * Tubal ligation
     * Partner's vasectomy
   * Examples of additional effective methods:

     * Male condom
     * Diaphragm
     * Cervical Cap
8. Subject has a body mass index (BMI) ≥ 18 and ≤ 33 kg/m2 at screening.
9. Protocol-specified clinical laboratory safety test results should be within the reference range of the clinical laboratory being used by the study site at screening and at baseline (Day -1).
10. Subject is afebrile, with supine systolic blood pressure (BP) ≥ 100 and ≤ 140 mmHg, supine diastolic BP ≥ 50 and ≤ 90 mmHg, and resting pulse rate ≥ 40 and ≤ 110 bpm at screening and Day -1.
11. Subject has a normal or clinically acceptable 12-lead electrocardiogram (ECG), with a QTcF value ≤ 430 msec, at screening and Day -1.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Subject has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Subject has any condition including the presence of laboratory abnormalities, which places the subject or other study participants at unacceptable risk if he were to participate in the study.
3. Subject has a past or current history of any condition affecting calcium homeostasis including, but not limited to: hypocalcemia, parathyroid disorders, vitamin D level lower than 20 ng/mL, disorders of phosphate or magnesium metabolism. The Investigator should contact the Sponsor for questions on any disorders that may be related to calcium homeostasis. Subjects with vitamin D levels < 30 ng/mL are not permitted to serve as sentinel subjects or alternates for the sentinel subjects.
4. Subject has a history of prior infusion reactions, anaphylactic reactions, or anaphylactoid reactions to any medication regardless of severity.
5. Subject participated in a radiolabeled drug study, where exposures either are known or unknown to the Investigator, within the previous 12 months prior to Day -1. The total 12-month exposure from this study and a maximum of 2 other previous studies within 4 to 12 months of this study will be within the CFR recommended levels considered safe, per US Title 21 CFR 361.1: less than 5,000 mrem whole body annual exposure, with consideration given to the half-lives of the previous radiolabeled study drugs received.
6. Subject was exposed to significant radiation (eg, serial X-ray or computed tomography scans, barium meal, current employment in a job requiring radiation exposure monitoring) within 12 months prior to Day -1. All questions regarding this criterion should be discussed with the Sponsor.
7. History of less than 1 to 2 bowel movements per day.
8. Subject is unable to take calcium citrate, vitamin D3, Dulcolax®, acetaminophen or diphenhydramine because of allergy or other intolerance.
9. Subject has any condition that confounds the ability to interpret data from the study. The Investigator should contact the Sponsor for questions about eligibility based on this criterion.
10. Subject was exposed to an investigational drug (new chemical entity) within 30 days prior to dosing, or 5 half-lives of that investigational drug, if known (whichever is longer).
11. Subject has used any prescribed systemic or topical medication (including but not limited to analgesics, anesthetics, etc) within 14 days or 5 half-lives of that medication, whichever is longer, prior to dosing.
12. Subject has used any non-prescribed systemic or topical medication (including vitamin/mineral supplements and herbal medicines) within 7 days prior to dosing.
13. Subject has used cytochrome P (CYP) 450 inducers and/or inhibitors (including St. John's Wort) within 30 days prior to dosing. The Indiana University "Cytochrome P450 Drug Interaction Table" should be utilized to determine inducers and/or inhibitors of CYP (http://medicine.iupui.edu/clinpharm/ddis/table.aspx).
14. Subject has any surgical or medical conditions possibly affecting drug absorption, distribution, metabolism, and excretion, eg, bariatric procedure. Note: prior appendectomy is acceptable, but prior cholecystectomy would result in exclusion from the study.
15. Subject donated blood or plasma within 8 weeks prior to dosing to a blood bank or blood donation center.
16. Subject has a history of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual [DSM]) within 2 years prior to dosing, or positive drug test reflecting consumption of illicit drugs.
17. Subject has a history of alcohol abuse (as defined by the current version of the DSM) within 2 years prior to dosing, or positive alcohol test.
18. Subject is known to have serum hepatitis or known to be a carrier of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (HCV Ab), or have a positive result to the test for human immunodeficiency virus (HIV) antibodies at screening.

    a. Note: Subjects who received hepatitis B vaccination and who test positive for hepatitis B surface antibody and negative for both hepatitis B surface antigen and hepatitis B core antibody remain eligible for study participation.
19. Subject smokes > 10 cigarettes per day, or equivalent in other tobacco products including eCigarettes or vapes (self-reported).
20. Subject has received immunization with a live or live attenuated vaccine within 2 months prior to dosing or is planning to receive immunization with a live or live attenuated vaccine for 2 months following dosing.
21. Subject is part of the study site personnel or a family member of the study site staff.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - Total [14C]- radioactivity (RA) | pre-dose to 240 hours post-dose
  Total [14C]-RA in whole blood, plasma, urine, and feces will be measured via LC-AMS
Pharmacokinetics - Cumulative excretion of total [14C]-RA | pre-dose to 240 hours post-dose
  Total RA recovery will be computed as the sum of the cumulative excretion (as % dose) in urine and feces.
Pharmacokinetics - Total [14C]-RA whole blood-to-plasma ratios | pre-dose to 120 hours post-dose
  Ratio of total RA recovery in whole blood compared to in plasma
Pharmacokinetics - Cmax | pre-dose to 240 hours post-dose
  Observed maximum concentration
Pharmacokinetics - AUC | pre-dose to 240 hours post-dose
  Area under the concentration
Pharmacokinetics - Tmax | pre-dose to 240 hours post-dose
  Time to Cmax.
Pharmacokinetics - t1/2 | pre-dose to 240 hours post-dose
  Terminal elimination half-life

SECONDARY OUTCOMES:
Adverse Events (AEs) | From the time of informed consent until 28 days after the last dose of study drug.
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values, regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a preexisting condition) should be considered an AE.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Covance Clinical Research Unit Inc., Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/